CLINICAL TRIAL: NCT03648099
Title: Effect of Labor Dance and Music on Labor Pain and Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, İlknur Münevver Gönenç, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Study of Labor Dance and Music
Record Dates: First submitted 2018-08-17; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Labor Pain; Fear of Childbirth
Keywords: Labor Pain; Labor dance; Music; Fear of childbirth
MeSH Terms: conditions — Labor Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: a single-blind randomized controlled intervention trial
Who Masked: Care Provider
Masking Description: In order to avoid bias in assessing pain and fear, three midwives who were not involved in the study team, who worked in the hospital where the study was carried out and who did not know the groups of the participants administered the scales. The midwives who were involved in data collection during the study were trained by the researchers on the use of data collection tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor Dance and music groups (Experimental): 1. Labor Dance; The pregnant women performed labor dance when the cervical dilatation reached 4-5 cm. The dance was performed in the company of music played through headphones.
  2. The pregnant women listened to music for 30 minutes when the cervical dilatation reached 4-5 cm. They took any position they wanted while listening to music.
  Interventions: Behavioral: Labor dance; Behavioral: Music
- Control group (No Intervention): The control group: No intervention was made to relieve the labor pain and reduce the fear of childbirth in the control group of the study. They were administered routine hospital applications.

INTERVENTIONS:
Behavioral: Labor dance — The dance group which involved pregnant women who performed the labor dance
  Arms: Labor Dance and music groups
Behavioral: Music — The music group involving pregnant women who were exposed to music.
  Arms: Labor Dance and music groups

SUMMARY:
The study was conducted to investigate the effect of labor dance and music used during the active phase of labor on labor pain and fear of childbirth. The study was designed as a single-blind randomized controlled intervention trial. The participants included in sample are taken into 3 groups (totally 93 participants). A total of 93 individuals, 31 of whom were in the dance group (D), 30 in the music group (M), and 32 in the control group (C), were included in the survey. Data were collected between 15 February 2018 and 15 June 2018 by means of a Personal Information Form, the Labor Monitoring Form, the Visual Analogue Scale (VAS), and version A of the Wijma Delivery Expectancy Questionnaire (W-DEQA).

DETAILED DESCRIPTION:
The study was designed as a single-blind randomized controlled trial with one control and two intervention groups. The aim of the study was to investigate the effect of labor dance and music used in the active phase of labor on perceived labor pain and fear of childbirth.

The hypotheses of our study are as follows:

H1: The labor dance used in the active phase of labor has an effect on reducing the perceived labor pain.

H2: The music used in the active phase of labor has an effect on reducing the perceived labor pain.

H3: The labor dance used in the active phase of labor has an effect on reducing the fear of childbirth.

H4: The music used in the active phase of labor has an effect on reducing the fear of childbirth.

H5: The labor dance is a more effective method in reducing the labor pain perceived in the active phase of labor compared to music.

H6: The labor dance is a more effective method in reducing the fear of childbirth in the active phase of labor compared to music.

There were three groups in the study: the dance group (D) which involved pregnant women who performed the labor dance; the music group (M) involving pregnant women who were exposed to music; the control group (C) which included pregnant women who were administered routine hospital practices. The sampling included pregnant women who met the inclusion criteria and agreed to participate in the study. D; The pregnant women performed labor dance when the cervical dilatation reached 4-5 cm. The dance was performed in the company of music played through headphones. The labor dance lasted 30 minutes. M; The pregnant women listened to music for 30 minutes when the cervical dilatation reached 4-5 cm. They took any position they wanted while listening to music. C; No intervention was made to relieve the labor pain and reduce the fear of childbirth in the control group of the study. They were administered routine hospital applications.The study data were collected using a Personal Information Form, the Labor Monitoring Form, the Visual Analogue Scale (VAS), and version A of the Wijma Delivery Expectancy Questionnaire (W-DEQA). After the pregnant women were randomly assigned to groups, the personal information form was filled in. The perceived pain and fear of the pregnant women in group D and group M were measured and recorded prior to the intervention (when cervical dilatation reached 4-5 cm). A 30-minute long intervention was administered in groups D and M. The pain and fear measurements were repeated soon after the intervention, 30 minutes and 60 minutes after the intervention. On the other hand, the pain and fear assessments in the control group were made when the cervical dilatation reached 4-5 cm. The assessment of the perceived pain and fear in controls who were administered routine hospital practices were repeated 30 minutes after the first measurement, after 60 minutes, and after 90 minutes .

ELIGIBILITY:
Inclusion Criteria:

1. An indication for vaginal delivery
2. Primipara
3. Cervical dilatation of 3 cm or over
4. Full-term pregnancy (38-42 gestational weeks)
5. Single healthy fetus in vertex position
6. No complication that can cause dystocia in labor (such as contraction anomalies, birth object, birth canal associated dystocia, maternal psychology associated dystocia)
7. Not using analgesia and anesthesia during the first phase of the labor
8. Having no physical disability to dance
9. Having no difficulty to take upright position and move
10. Having no communication problem.

Exclusion Criteria:

1. Giving up participating in the study
2. Abnormal changes in fetal heartbeat
3. Emergence of an unexpected complication in the pregnant woman or the fetus 4) Taking analgesics and anesthesia

5) Incomplete intervention and follow-up due to rapid labor 6) Being taken to C/S before the completion of the intervention and follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Score, | Baseline
  The perceived pain pregnant women in groups were measured and recorded prior to the intervention (when cervical dilatation reached 4-5 cm).
  Assessed the labor pain level with Visual Analogue Scale score. This is a 10 cm scale which is labeled "no pain" at one end and "severe pain" at the other end. (0=no pain; 10= pain as bad as can be). Increasing scores indicate women's labor pain.

SECONDARY OUTCOMES:
Version A of the Wijma Delivery Expectancy Questionnaire Score | Baseline
  The fear pregnant women in groups were measured and recorded prior to the intervention (when cervical dilatation reached 4-5 cm). Assessed childbirth of fear with version A of the Wijma Delivery Expectancy. Questionnaire score. The minimum and maximum scores that can be obtained from the scale range between 0 and 165. Increasing scores indicate women's fear of childbirth.
Recurrence of Fear of Childbirth | 30 minutes, 60 minutes and 90 minutes
  A 30-minute long intervention was administered in groups Dance and Music. The fear measurements were repeated soon after the intervention, 30 minutes and 60 minutes after the intervention. Assessed childbirth of fear with version A of the Wijma Delivery Expectancy. Questionnaire score. The minimum and maximum scores that can be obtained from the scale range between 0 and 165. Increasing scores indicate women's fear of childbirth.
Recurrence of perceived pain | 30 minutes, 60 minutes and 90 minutes
  Measurements were repeated 30 minutes after the first measurement, after 60 minutes, and after 90 minutes.
  Assessed the labor pain level with Visual Analogue Scale score. This is a 10 cm scale which is labeled "no pain" at one end and "severe pain" at the other end. (0=no pain; 10= pain as bad as can be). Increasing scores indicate women's labor pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdul-Sattar Khudhur Ali S, Mirkhan Ahmed H. Effect of Change in Position and Back Massage on Pain Perception during First Stage of Labor. Pain Manag Nurs. 2018 Jun;19(3):288-294. doi: 10.1016/j.pmn.2018.01.006. Epub 2018 Apr 19. PMID 29680213
- [Result] Whitburn LY, Jones LE, Davey MA, Small R. Women's experiences of labour pain and the role of the mind: an exploratory study. Midwifery. 2014 Sep;30(9):1029-35. doi: 10.1016/j.midw.2014.04.005. Epub 2014 Apr 30. PMID 24820004
- [Result] Simavli S, Kaygusuz I, Gumus I, Usluogullari B, Yildirim M, Kafali H. Effect of music therapy during vaginal delivery on postpartum pain relief and mental health. J Affect Disord. 2014 Mar;156:194-9. doi: 10.1016/j.jad.2013.12.027. Epub 2013 Dec 28. PMID 24411681
- [Result] Masoudi Z, Akbarzadeh M, Vaziri F, Zare N, Ramzi M. The effects of decreasing maternal anxiety on fetal oxygenation and nucleated red blood cells count in the cord blood. Iran J Pediatr. 2014 Jun;24(3):285-92. PMID 25562022
- [Result] Gokyildiz Surucu S, Ozturk M, Avcibay Vurgec B, Alan S, Akbas M. The effect of music on pain and anxiety of women during labour on first time pregnancy: A study from Turkey. Complement Ther Clin Pract. 2018 Feb;30:96-102. doi: 10.1016/j.ctcp.2017.12.015. Epub 2017 Dec 19. PMID 29389487
- [Result] Abdolahian S, Ghavi F, Abdollahifard S, Sheikhan F. Effect of dance labor on the management of active phase labor pain & clients' satisfaction: a randomized controlled trial study. Glob J Health Sci. 2014 Mar 30;6(3):219-26. doi: 10.5539/gjhs.v6n3p219. PMID 24762366
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203